CLINICAL TRIAL: NCT04344587
Title: Awake Prone Position for Early Hypoxemia in COVID-19
Acronym: APPEX-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: H-40070
Record Dates: First submitted 2020-04-08; First posted 2020-04-14 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: COVID-19
Keywords: Prone position; Coronavirus; Inhalation oxygen therapy; Pragmatic Clinical Tria; Hypoxia
MeSH Terms: conditions — COVID-19; Coronavirus Infections; Hypoxia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Participants in the intervention arm will receive a text message on their smartphones linking to the Qualtrics intervention website
  Interventions: Other: Self-prone position recommendation
- Usual care group (Active Comparator): Participants in the usual care arm will receive a text message on their smartphone linking to the Qualtrics usual care website
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Self-prone position recommendation — The Qualtrics self-prone position recommendation intervention website will include the following sections:
  1. Welcome message
  2. Educational review of the potential benefits of prone positioning
  3. How-To guide to safely "prone" in a hospital bed
  4. A recommendation to "prone" while lying in bed (4 times for 1-2 hours each during the day and at night every 24 hours).
  5. A reminder to keep track of the time spent in 1) prone position, 2) lying flat on back, 3) lying on side, 4) sitting up, and 5) standing or walking
  Arms: Intervention group
Other: Usual care — The Qualtrics usual care website will include the following sections:
  1. Welcome message
  2. A reminder to keep track of the time spent in 1) prone position, 2) lying flat on back, 3) lying on side, 4) sitting up, and 5) standing or walking
  Arms: Usual care group

SUMMARY:
Prone positioning is a well studied and validated treatment for severe acute respiratory distress syndrome (ARDS), however there are no randomized studies on the use of prone positioning in the non-intubated patient. It is unknown if this intervention would be helpful in preventing further respiratory deterioration in terms of increasing supplemental oxygen requirements, endotracheal intubation, and ICU admission.

The Awake Prone Position for Early hypoxemia in COVID-19 (APPEX-19) Study is a pragmatic adaptive randomized controlled unblinded trial. APPEX-19 randomizes non-ICU patients with COVID-19 or who are under evaluation for COVID-19 to lie in a prone position (i.e, with their stomach and chest facing down) or to usual care.

DETAILED DESCRIPTION:
The purpose of this multi-site trial is to investigate the use of prone positioning in SARS-CoV-2 infected patients who are not intubated. The APPEX-19 study is a pragmatic adaptive randomized controlled unblinded trial. The study compares a smartphone tool that recommends non-ICU patients with COVID-19 or who are under evaluation for COVID-19 to lie in a prone position (i.e, with their stomach and chest facing down) to usual care.

Participants who are assigned to the intervention arm will receive a text message containing a link to an online website that reviews how to safely self-prone position and a recommendation to self-prone position 4 times for 1-2 hours each during the day and at night every 24 hours. Participants will also receive twice daily reminders to self-prone using the same smartphone platform.

All participants will receive twice daily Qualtrics online surveys to answer questions about which body positions they used in bed and their level of comfort and shortness of breath. Participants will receive these twice daily text messages until they are discharged, until they are transferred to the ICU, until they die, until their lung function declines, or until 14 days pass since enrollment. Thus, most participants will receive twice daily text messages for about 1 week; it is expected that almost all patients will receive twice daily text messages for no longer than 14 days. Medical charts will be reviewed daily to track routine clinical data to determine outcomes.

Boston Medical Center (BMC) / Boston University will be one of the 16 sites and the data coordinating center for this multisite trial. The unique design of the study means that if evidence accumulates that one treatment is better than the other, more participants will be chosen to receive the prone position intervention that works over time. Thus, the trial will both show what works, implement what works, and make sure that the most participants receive the treatment that works.

ELIGIBILITY:
Inclusion Criteria:

* Assigned to or admitted to a COVID-19 ward team at a participating site (these teams only admit patients who are under investigation for COVID-19 or who have confirmed COVID-19 infection) via the emergency department (ED) within the last 24 hours
* Have access to their own functioning smartphone in the hospital room
* English or Spanish-speaking
* Ability to read simple instructions and answer simple written questions

Exclusion Criteria:

Baseline patient factors

* Inability to operate the hospital bed
* Inability to lie flat comfortably
* Inability to lie flat without shortness of breath
* Inability to turn over independently

Medical comorbidities

* Hemoptysis in the last 2 days
* Prior lung transplant
* Dementia

Acute issues

* Deep venous thrombosis treated for less than 2 days
* Unstable spine, femur, or pelvic fractures
* Mean arterial pressure lower than 65 mmHg
* Receiving ≥6 liters per minute of supplemental oxygen via nasal cannula, nasal pendant, or shovel mask
* Receiving supplemental oxygen via more aggressive methods (e.g. Venturi mask or non-rebreather mask)

Recent interventions

* Chest tube in place
* Tracheal surgery or sternotomy during the previous 15 days
* Serious facial trauma or facial surgery during the previous 15 days
* Cardiac pacemaker inserted in the last 2 days

Other

* Pregnancy
* Comfort measures only status
* Prisoner

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 305 (Actual)
Dates: Start 2020-04-23 (Actual); Primary Completion 2021-05-07 (Actual); Study Completion 2021-05-07 (Actual)

PRIMARY OUTCOMES:
Change in respiratory status | up to 30 days
  Change in respiratory status will be defined as:1) admission to the ICU and/or a 2) an increase in supplemental oxygen delivery (defined as an increase in oxygen delivery rate of ≥2 liter per minute compared to the oxygen delivery rate at the time of intervention or usual care text message that is sustained for ≥12 or more hours OR the switch to an oxygen delivery method that increases the level of supplemental oxygen.

SECONDARY OUTCOMES:
Length of time participant spends in the prone position | up to 30 days
  Length of time in the prone position will be assessed from the smartphone survey and measured in categories of no time, up to 6 hours, 6 hours to 11 hours, 12 hours or more.
Length of time participant spends in the supine position | up to 30 days
  Length of time in the supine/lying on back position will be assessed from the smartphone survey and measured in categories of no time, up to 6 hours, 6 hours to 11 hours, 12 hours or more.
Length of time participant spends lying on side | up to 30 days
  Length of time lying on side will be assessed from the smartphone survey and measured in categories of no time, up to 6 hours, 6 hours to 11 hours, 12 hours or more.
Length of time participant spends sitting up | up to 30 days
  Length of time sitting up will be assessed from the smartphone survey and measured in categories of no time, up to 6 hours, 6 hours to 11 hours, 12 hours or more.
Length of time participant spends standing or walking | up to 30 days
  Length of time standing or walking will be assessed from the smartphone survey and measured in categories of no time, up to 6 hours, 6 hours to 11 hours, 12 hours or more.
Dyspnea or difficult/labored breathing | up to 30 days
  Dyspnea will be assessed by the modified Borg Dyspnea Score (10-point ordinal scale) from 1= nothing at all to 10= maximal. Higher scores indicate more dyspnea.
Discomfort with proning | up to 30 days
  Discomfort with proning (4-point ordinal scale: very comfortable, somewhat comfortable, somewhat uncomfortable, very uncomfortable)
Length of hospital stay | up to 30 days
  Total number of days hospitalized will be abstracted from the electronic medical record.
Invasive mechanical ventilation | up to 30 days
  Invasive mechanical ventilation will be abstracted from the electronic medical record.
Loss of IV access as a consequence of turning in bed | up to 30 days
  Loss of IV access as a consequence of turning in bed will be reported by participant using monitoring surveys
Acute respiratory distress syndrome (ARDS) diagnosis | up to 30 days
  ARDS diagnosis will be abstracted from the electronic medical record
Hospital mortality | up to 30 days
  Hospital mortality will be abstracted from the electronic medical record

CONTACTS AND LOCATIONS:
Overall Officials: Allan J Walkey, MD, Study Director — Boston University
Locations (13):
- United States (12):
  - Long Beach Medical Center - MemorialCare, Long Beach, California
  - Alvarado Hospital, San Diego, California
  - St. Joseph's Hospital National Jewish Health, Denver, Colorado
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Piedmont Atlanta, Atlanta, Georgia
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Boston Medical Center, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Creighton University, Omaha, Nebraska
  - Michael E. DeBakey Veteran Affairs Medical Center, Houston, Texas
  - VCU Medical Center, Richmond, Virginia
- Hospital Universitario La Paz, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Garcia MA, Rampon GL, Doros G, Jia S, Jagan N, Gillmeyer K, Berical A, Hudspeth J, Ieong M, Modzelewski KL, Schechter-Perkins EM, Ross CS, Rucci JM, Simpson S, Walkey AJ, Bosch NA. Rationale and Design of the Awake Prone Position for Early Hypoxemia in COVID-19 Study Protocol: A Clinical Trial. Ann Am Thorac Soc. 2021 Sep;18(9):1560-1566. doi: 10.1513/AnnalsATS.202009-1124SD. PMID 33647225
- [Derived] Rampon G, Jia S, Agrawal R, Arnold N, Martin-Quiromicrons A, Fischer EA, Malatack J, Jagan N, Sergew A, Case AH, Miller K, Tanios M, Doros G, Ross CS, Garcia MA, Gillmeyer KR, Griffiths NG, Jandali B, Modzelewski KL, Rucci JM, Simpson SQ, Walkey AJ, Bosch NA. Smartphone-Guided Self-prone Positioning vs Usual Care in Nonintubated Hospital Ward Patients With COVID-19: A Pragmatic Randomized Clinical Trial. Chest. 2022 Oct;162(4):782-791. doi: 10.1016/j.chest.2022.05.009. Epub 2022 May 18. PMID 35597286